CLINICAL TRIAL: NCT00067366
Title: Brief Focused Treatment for TMD: Mechanisms of Action
Brief Title: Brief Treatment for Temporomandibular Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Responsible Party: Principal Investigator, Mark Litt, Professor, UConn Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDCR-14607
Record Dates: First submitted 2003-08-15; First posted 2003-08-19 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Temporomandibular Joint Syndrome; Myofascial Pain Dysfunction Syndrome; Orofacial Pain
MeSH Terms: conditions — Temporomandibular Joint Dysfunction Syndrome; Fibromyalgia; Facial Pain

ARMS (2):
- Coping Skills Training (Experimental): manualized coping skills training delivered along with conservative care
  Interventions: Behavioral: Cognitive-Behavioral treatment
- Standard Care (Active Comparator): Attention and life counseling added to Standard conservative care
  Interventions: Behavioral: Attention and lifestyle counseling

INTERVENTIONS:
Behavioral: Cognitive-Behavioral treatment — Cognitive-Behavioral skills training for chronic pain
  Arms: Coping Skills Training
Behavioral: Attention and lifestyle counseling — Attention and lifestyle counseling added to Standard Care
  Arms: Standard Care

SUMMARY:
Temporomandibular Disorder (TMD) is a widespread chronic pain condition. Successful psychosocial treatments for TMD have been developed, but the mechanisms by which these treatments achieve their effects are not well known. The goal of this project is to evaluate the possible mechanisms responsible for treatment gains in TMD treatment.

DETAILED DESCRIPTION:
TMD is a widespread chronic pain condition. Successful psychosocial treatments for TMD have been developed, but the mechanisms by which these treatments achieve their effects are not well known. The goal of this project is to evaluate the possible mechanisms responsible for treatment gains in TMD treatment. Men and women (N=106) with complaints of chronic facial pain for at least 3 months' duration will be recruited from the University Dental Clinics and from the community via advertisements and randomly assigned to either a Standard Conservative Treatment (STD) employing an intraoral splint plus anti-inflammatory agents, or to a Standard Treatment + Cognitive-Behavioral Treatment Program (STD+CBT), that will include standard treatment but also focus on changing self-efficacy and decreasing catastrophization. Both treatments will entail 6 clinic visits. Dispositional and situational variables derived from a comprehensive model of pain coping will be measured before and after treatment. The situational variables, including coping responses, mood states, situational appraisals and self-efficacy, will be measured in an experience sampling paradigm four times daily using a hand-held computer. This will be done to minimize retrospective biases that may have hampered earlier studies of treatment process. Dependent variables will be self-report measures of distress, pain, and interference with activities, as well as blood plasma levels of cortisol and selected cytokines, measured at the end of the 6-week treatment period, and at follow-up points thereafter up to a 12-month follow-up. It is expected that the STD+CBT treatment will result in measurable changes in constructs such as self-efficacy and catastrophization, and that these changes will be related to improved outcomes compared to the STD controls. It is also expected that outcome differences between groups will be associated with changes in inflammatory mediators (cytokine levels). Finally, it is suggested that changes in situational treatment process variables will be associated with changes in cytokine levels. The results may indicate the true active mechanisms of successful TMD treatment. If these mechanisms can be successfully identified it would have important implications for the development of more effective treatment programs.

ELIGIBILITY:
Inclusion Criteria:

* Complaining of chronic TM-related pain for at least 3 months
* Positive Axis I diagnosis on the Research Diagnostic Criteria (RDC) for temporomandibular disorders (positive on at least one Group), and may have no contraindications to TMD treatment
* Fluency in English

Exclusion Criteria:

* No previous surgery for treatment of TMD pain
* No history of rheumatoid disease
* No extensive anatomical destruction or deterioration of the TM joint
* Not diagnosed as having pain of neuropathic or odontogenic origin
* Not carrying a diagnosis of psychosis
* No current treatment for depression
* Not taking narcotic pain medication
* Not pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2003-10; Primary Completion 2008-10 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Pain | Every 3 months out to 12 months
  Multidimensional pain ratings collected in person every 3 months
Pain-related interference with functioning | every 3 months out to 12 months
  Multidimensional function ratings collected in person every 3 months
Depressive symptoms | Every 3 months out to 12 months
  CES-D depressive symtpoms scale administered in perosn every 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Litt, Ph.D., Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States